CLINICAL TRIAL: NCT06300658
Title: Stellate Ganglion Block for Preserving Arteriovenous Fistula in Hemodialysis Patients Undergoing Major Lower Limb Orthopedic Surgery: A Randomized Controlled Trial
Brief Title: Stellate Ganglion Block for Preserving Arteriovenous Fistula in Hemodialysis Patients Undergoing Major Lower Limb Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Ayman Mohamady Eldemrdash, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Aswan University, Egypt, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 900/2/24
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-03

CONDITIONS: Stellate Ganglion Block; Arteriovenous Fistula; Hemodialysis; Major Lower Limb Orthopedic Surgery
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stellate ganglion blockade (Experimental): Patient will receive preemptive stellate ganglion blockade (SGB) just before spinal anesthesia.
  Interventions: Drug: Stellate ganglion block
- Control group (No Intervention): Patient will not receive preemptive stellate ganglion blockade (SGB).

INTERVENTIONS:
Drug: Stellate ganglion block — Patient will receive preemptive stellate ganglion block (SGB) just before spinal anesthesia.
  Arms: Stellate ganglion blockade

SUMMARY:
The aim of this study is to evaluate the role of stellate ganglion blockade (SGB) for preserving arteriovenous fistula in hemodialysis patients undergoing major lower limb orthopedic surgery.

DETAILED DESCRIPTION:
The best way for dialysis in chronic renal failure (CRF) patients with consideration of feasibility, rate of infection, and patency is hemodialysis by using native access by using arteriovenous fistula (AVF).

Altered calcium and phosphor metabolism in CRF patients would also increase vascular reactivity. Stellate ganglion blockade (SGB) has been used for several years for both diagnosis and treatment of circulatory problems in upper extremity. Recently preemptive SGB has been used in prevention of radial artery spasm in coronary artery patients.

SGB increases blood flow and decrease vascular resistance in the arm. SGB prevents or ameliorates the reactivity of the muscular layer of the RA in response to both surgical manipulation during harvesting the artery and to the potent vasoconstrictor mediators released during surgery

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status III.
* Chronic renal failure (CRF) patients.
* Undergoing major lower limb orthopedic surgery.

Exclusion Criteria:

* Psychiatric disorders.
* History of substance abuse.
* Ipsilateral brachial and radial artery stenosis.
* Allergy to local anesthetics.
* Cardiovascular and respiratory disorders.
* Coagulopathy.
* Use of vasoactive medications.
* Obesity (body mass index >30 kg/m2).
* Smoking.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Fistula flow rate | 7th day postoperatively
  Flow rate will be measured on the first day postoperative then on the 7th day.

SECONDARY OUTCOMES:
Peak systolic velocity (PSV) | 7th day postoperatively
  Peak systolic velocity (PSV) will be measured from radial artery 2 cm. proximal to fistula site, on the first day postoperative then on the 7th day.
End diastolic velocity (EDV) | 7th day postoperatively
  End diastolic velocity (EDV) will be measured from radial artery 2 cm. proximal to fistula site, on the first day postoperative then on the 7th day.
Incidence of failure | 7th day postoperatively
  Incidence of failure will be measured on the first day postoperative then on the 7th day.
Adverse effects | 7th day postoperatively
  Postoperative adverse reactions such as hematoma, infection, thrombosis, bleeding, and pitosis will be recorded in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Eldemrdash AM, Hammad SS, Hemaida TS, Dardeer TT, Mohsen AA, Fathy AK, Shams GH. Stellate ganglion block for preserving arteriovenous fistula in hemodialysis patients undergoing major lower limb orthopedic surgeries: randomized control trial. BMC Anesthesiol. 2025 May 31;25(1):277. doi: 10.1186/s12871-025-03150-7. PMID 40450242